CLINICAL TRIAL: NCT01509989
Title: International Prospective Study on Adherence to Treatment in Patients With Active Systemic Lupus Erythematosus
Acronym: Adherence-SLE
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: Record2012
Record Dates: First submitted 2011-12-01; First posted 2012-01-13 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Adherence; Compliance; Systemic Lupus Erythematosus; Hydroxychloroquine; Blood monitoring; Flares
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Patient Compliance

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The treatment of systemic lupus erythematosus (SLE) may change in the future due to the availability of new biological treatments, especially monoclonal antibodies in patients with active disease. However, one of the main causes of treatment failure in SLE is the lack of treatment adherence since "drugs don't work in patients who don't take them." Hydroxychloroquine (HCQ-Plaquenil) has a long terminal elimination half- life, and investigators have demonstrated that patients who do not take HCQ for a long time have undetectable or very-low blood HCQ concentrations (< 200 ng/ml). The rate of severe non-adherence was 7% in a cohort of 203 patients and was even higher in patients with active disease: 8 out of 35 (23%) in patients with a SLEDAI ≥6 and 6 out of 20 (30%) in patients with a SLEDAI ≥12.

Investigators will evaluate the importance of non-adherence to the treatment in a large population of SLE patients with active disease. This will be done with blood HCQ monitoring in a translational multicentric prospective study.

DETAILED DESCRIPTION:
This international multicentric prospective study is an observational study that will include consecutive SLE patients treated with HCQ and with SLE flare (defined by the SELENA-SLEDAI flare composite). The study will only require the sampling of 1 vial of whole blood for the dosage of HCQ (that would be centralized and performed in PITIE-SALPETRIERE Hospital at the completion of the study). The patients and the physicians will also have adherence self-questionnaires to complete, and the physicians will complete a patient data sheet.

The end points are adherence of the treatment in the whole group, and subgroups, adherence according to the severity of SLE, and the relationship between patient's questionnaires, physician evaluation of adherence and blood HCQ dosage.

If investigators confirm their previous data, this study might demonstrate that a significant proportion of patient candidates for treatment escalation are in fact nonadherent to the treatment. It might further demonstrate the interest of HCQ concentrations monitoring, both in "real life" and in therapeutic study in SLE as it may avoid unnecessary, expensive or even hazardous regimen escalation.

ELIGIBILITY:
Inclusion criteria :

* History of meeting 4 American College of Rheumatology (ACR) criteria for systemic lupus erythematosus including a positive test for antinuclear antibodies,
* SLE flare defined by the SELENA-SLEDAI flare composite
* Treatment with HCQ for at least 2 months with a daily dosage > or equal to 200 mg/day.

Exclusion criteria :

* Patients who are not able to take their medications (notably patients with repeated vomiting and patients who are not allowed to take oral medications)

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Active Systemic Lupus Erythematosus (see eligibility criteria)
Sampling Method: Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Adherence to the treatment in the whole group. | participants will be followed for the duration of hospital stay, an expected average of 1
  The end points are adherence of the treatment in the whole group(defined by very low blood HCQ concentration)

SECONDARY OUTCOMES:
Secondary outcome | up to 3 weeks
  Adherence according to central nervous system, to pregnancy, to the severity of SLE, to the center and the country.
  Adherence in the group of patients fulfilling the eligibility criteria of studies on monoclonal antibodies, The relationship between patients questionnaires, physician evaluation of adherence and blood HCQ dosage Interest of MASRI and Morisky questionnaires in the prediction of non-adherence Factors associated with poor adherence
  The socio-economic aspect of blood HCQ concentration measurement Pharmacokinetics studies on HCQ, with comparison to another cohort

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Costedoat-Chalumeau, MD, Principal Investigator — Service de Médecine Interne, Hopital Cochin, 27, rue du Faubourg St Jacques, 75014 Paris, France. Email : nathalie.costedoat@gmail.com; Michelle Petri, MD, Principal Investigator — Dept of Rheumatology, 1830 Building, Suite 7500. Email: mpetri@jhmi.edu; Jill Buyon, MD, Principal Investigator — 560 First avenue, TCH-407, New York-NY 10016. Email: jill.buyon@nyumc.org; Ann Clarke, MD, Principal Investigator — Lupus Clinic, Montreal General Hospital, Room A6163, 1650 Cedar Ave, Montreal, Quebec, Canada, H3G 1A4. Email: ann.clarke@mcgill.ca; Frederic Houssiau, MD, Principal Investigator — Rheumatology Unit, Internal Medicine Department, Cliniques universitaires Saint-Luc, Université catholique de Louvain,Bruxelles, Belgium. Email: Frederic.Houssiau@uclouvain.be; Guillermo Ruiz-Irastorza, MD, Principal Investigator — Autoimmune Disease Research Unit, Internal Medicine Department,Hospital de Cruces, University of the Basque Country, Barakaldo, Spain. Email: r.irastorza@euskaltel.net; Ricard Cervera, MD, Principal Investigator — Department of Autoimmune Diseases, Hospital Clínic, rcervera@clinic.ub.es Barcelona, Catalonia, Spain. Email: rcervera@clinic.ub.es; David Isenberg, MD, Principal Investigator — Department Inflammation, UCL Division of Medicine, Room 331 The Windeyer Building, 46 Cleveland Street, London, England. Email: d.isenberg@ucl.ac.uk; Yehuda Shoenfeld, MD, Principal Investigator — Zabludowicz Center for Autoimmune Diseases, Sheba Medical Center, Tel-Hashomer 52621, Israel. Email: shoenfel@post.tau.ac.il; Ronald F. van Vollenhoven, MD, Principal Investigator — Unit for Clinical Therapy Research, Inflammatory Diseases (ClinTRID), The Karolinska University Hospital, D10:0, Department of Rheumatology, 17176 Stockholm, Sweden. Email: Ronald.van.Vollenhoven@ki.se; Eric Hachulla, MD, Principal Investigator — Service de Médecine Interne, Hôpital Claude Huriez, 1, place Verdun, 59000 Lille. Email: ehachulla2@yahoo.fr; Jean-François Viallard, MD, Principal Investigator — Service de Médecine Interne, Hôpital Haut Lévêque, Centre François Magendie, 1, avenue Magellan, 33604 Pessac Cedex. Email: jean-francois.viallard@chu-bordeaux.fr; Loïc Guillevin, MD, Principal Investigator — Service de Médecine Interne, Hôpital Cochin, 27, rue du Faubourg Saint-Jacques, 75679 PARIS Cedex 14. Email: loic.guillevin@wanadoo.fr; Luc Mouthon, MD, Principal Investigator — Service de Médecine Interne, Hôpital Cochin, 27, rue du Faubourg Saint-Jacques, 75679 PARIS Cedex 14. Email: luc.mouthon@cch.aphp.fr; Veronique Leguern, MD, Principal Investigator — Service de Médecine Interne, Hôpital Cochin, 27, rue du Faubourg Saint-Jacques, 75679 PARIS Cedex 14.; Jean-Charles Piette, MD, Principal Investigator — Service de Médecine Interne, Hopital Pitié-Salpêtrière, 47-83 Boulevard de l'hôpital, 75013 Paris, France. Email: jcpiette@free.fr; Lionel Galicier, MD, Principal Investigator — Service Immuno Clinique; Anne Laure Fauchais, MD, Principal Investigator — Service de Médecine interne, Hôpital Dupuytren, 2, avenue Martin Luther King 87042 Limoges cedex; Holy Harifidy Bezanahrv, MD, Principal Investigator — Service de Médecine interne, Hôpital Dupuytren, 2, avenue Martin Luther King 87042 Limoges cedex; Christophe deligny, MD, Principal Investigator — Service de Médecine interne (3C), CHU de Martinique, Hôpital Pierre-Zobda-Quitman, CS 90631-97261 Fort de France cedex; Sandra Navarra, MD, Principal Investigator — University of Santo Tomas Hospital, España Boulevard, Sampaloc, Manila, Philippines
Locations (1):
- Hopital Cochin, Paris, France

REFERENCES:
- [Derived] Costedoat-Chalumeau N, Houssiau F, Izmirly P, Guern VL, Navarra S, Jolly M, Ruiz-Irastorza G, Baron G, Hachulla E, Agmon-Levin N, Shoenfeld Y, Dall'Ara F, Buyon J, Deligny C, Cervera R, Lazaro E, Bezanahary H, Leroux G, Morel N, Viallard JF, Pineau C, Galicier L, Vollenhoven RV, Tincani A, Nguyen H, Gondran G, Zahr N, Pouchot J, Piette JC, Petri M, Isenberg D. A Prospective International Study on Adherence to Treatment in 305 Patients With Flaring SLE: Assessment by Drug Levels and Self-Administered Questionnaires. Clin Pharmacol Ther. 2019 Aug;106(2):374-382. doi: 10.1002/cpt.1194. Epub 2018 Sep 2. PMID 30079582
- [Derived] Costedoat-Chalumeau N, Houssiau F, Izmirly P, Le Guern V, Navarra S, Jolly M, Ruiz-Irastorza G, Baron G, Hachulla E, Agmon-Levin N, Shoenfeld Y, Dall'Ara F, Buyon J, Deligny C, Cervera R, Lazaro E, Bezanahary H, Leroux G, Morel N, Viallard JF, Pineau C, Galicier L, Van Vollenhoven R, Tincani A, Nguyen H, Gondran G, Zahr N, Pouchot J, Piette JC, Petri M, Isenberg D. A Prospective International Study on Adherence to Treatment in 305 Patients With Flaring SLE: Assessment by Drug Levels and Self-Administered Questionnaires. Clin Pharmacol Ther. 2018 Jun;103(6):1074-1082. doi: 10.1002/cpt.885. Epub 2017 Nov 9. PMID 28925027